CLINICAL TRIAL: NCT01244672
Title: Trans-anal Hemorrhoidal Dearterialization (THD) vs. Hemorrhoidectomy for 3rd and 4th Degree Hemorrhoids in at Least Three Quadrants: A Prospective Randomized Control Pilot Study.
Brief Title: Trans-anal Hemorrhoidal Dearterialization (THD) vs. Hemorrhoidectomy
Acronym: THD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Roberto Bergamaschi, Professor and Chief, Division of colon and rectal surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106946
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; THD; Ferguson
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trans-anal dearterialization (Active Comparator): 24 patients were assigned to the Transanal hemorrhoidal dearterialization with mucopexy arm, which is a Doppler guided procedure for suture ligation of hemorrhidal arteries rather than excisional
  Interventions: Procedure: THD
- Ferguson (Active Comparator): 17 patients were randomized to Ferguson method, which is the operative gold standard for hemorrhoids. This is an excisional surgery.
  Interventions: Procedure: Ferguson

INTERVENTIONS:
Procedure: Ferguson — This is a modification of the Milligan-Morgan technique, whereby the incisions are totally or partially closed with absorbable running suture. A retractor is used to expose the hemorrhoidal tissue, which is then removed surgically. The remaining tissue is either sutured or is sealed through the coagulation effects of a surgical device.
  Arms: Ferguson
Procedure: THD — Transanal hemorrhoidal dearterialization will be performed using an endoscopic ultrasonic probe. Approximately 7-8 hemorrhoidal arteries will be ligated at 1, 3, 5, 7, 9, 11 o'clock position as previously described in the literature. The ligation will be performed using a vicryl suture. The ultrasonic probe locates the arterial signal.
  Arms: Trans-anal dearterialization

SUMMARY:
The purpose of this study is to compare the frequency and severity of postoperative( after surgery) pain between two surgical techniques for treating severe hemorrhoids. The two techniques are called: transanal hemorrhoidal dearterialization (THD) and standard surgical excision (removal) of the hemorrhoids

DETAILED DESCRIPTION:
The THD technique involves using ultrasound equipment to identify the arteries that are feeding blood into the hemorrhoids. Once located, stitches are placed around those arteries to cut off the blood supply to the hemorrhoids, which destroys them.

In the standard surgical excision technique, the hemorrhoids are removed by cutting them out with a scalpel.

Both techniques are widely used in many hospitals today. However, there have been no formal studies comparing the two techniques regarding outcomes, particularly regarding pain after the procedure. We plan to enroll 60 patients in this study here at Stony Brook; 30 patients will have THD and 30 will have the standard surgical excision of hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

Patients visiting colorectal outpatient office at Stony Book Medical Center, with the diagnosis of 3rd or 4th degree hemorrhoids requiring hemorrhoidectomy will be invited to participate in this study. The diagnosis of hemorrhoids will be established by a colorectal surgeon based on following criteria:

1. physical exam
2. anoscopy or proctoscopy

Exclusion Criteria:

1. first and second degree hemorrhoids
2. recurrent hemorrhoids after previous surgical treatment
3. history of HIV
4. history of inflammatory bowel disease
5. inability to give informed consent due to mental disability
6. age younger than 18
7. history of colon, rectal or anal cancer
8. thrombosed hemorrhoids
9. pregnant women
10. non English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 14 days
  Patient reports pain levels at 14 days post surgery

SECONDARY OUTCOMES:
complications | 30 days
  Complications involving hospital visit.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bergamaschi, MD, PhD, Principal Investigator — Stony Brook University Medical Center
Locations (1):
- State University Hospital Medical Center, Stony Brook, New York, United States